CLINICAL TRIAL: NCT04089579
Title: A Phase II Study of hCT-MSC, an Umbilical Cord-Derived Mesenchymal Stromal Cell Product, in Children With Autism Spectrum Disorder
Brief Title: hCT-MSC in Children With Autism Spectrum Disorder
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Marcus Foundation (Other); Cryo-Cell International (Unknown)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00113011; Pro00102894 (Other: Duke IRB)
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder; Stem cell; Mesenchymal Stromal Cells
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study is a phase II, prospective, randomized, blinded, cross over, clinical trial designed to assess the efficacy of intravenous dosing of hCT-MSC for improving social communication abilities in young children with ASD. All participants will ultimately be treated with hCT-MSC. Participants randomized to arm A will each receive a single intravenous dose of 6x106 hCT-MSC per kilogram at baseline, followed by a placebo infusion at six months. Participants randomized to arm B will each receive a placebo infusion at baseline, followed by an intravenous dose of 6x106 hCT-MSC per kilogram at six months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSC (Experimental): One dose of 6x10e6 cells/kg administered intravenously.
  Interventions: Biological: Cord Tissue Mesenchymal Stromal Cells
- Placebo Infusion (Placebo Comparator): Placebo infusion
  Interventions: Other: Placebo Infusion

INTERVENTIONS:
Biological: Cord Tissue Mesenchymal Stromal Cells — Human Umbilical Cord Tissue Derived Mesenchymal Stromal Cells (hCT-MSC), isolated and expanded from umbilical cord tissue from allogeneic unrelated donors. One dose of 6x10e6 cells/kg administered intravenously.
  Arms: MSC
Other: Placebo Infusion — Placebo comparative infusion
  Arms: Placebo Infusion

SUMMARY:
The purpose of this Phase II study is to determine the efficacy of human umbilical cord tissue-derived mesenchymal stromal cells (hCT-MSC) for improving social communication abilities in children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
The purpose of this double blinded Phase II study is to determine the efficacy of human umbilical cord tissue-derived mesencymal stromal cells (hCT-MSC), administered in two different dosing strategies, in children with autism spectrum disorder (ASD).

This study will be enrolling children with ASD, aging 4-11 years of age. Qualifying subjects will undergo neuropsychological evaluation, EEG testing, eye tracking, CVA assessments, and infusion of study product. Subjects will be randomized to one of two study arms; 1) a single infusion of 6.0x106 cells/Kg at baseline, followed by a blinded placebo infusion at six months or, 2) Placebo infusion at baseline, followed by an intravenous dose of 6x106 cells/Kg at six months.

The primary endpoint of this study is the change in social communication skill from baseline to six months. The potential risks associated with infusion of MSCs include a reaction to the product (rash, shortness of breath, wheezing, difficulty breathing, hypotension, swelling around the mouth, throat or eyes, tachycardia, diaphoresis), transmission of infection, and HLA sensitization.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 4 years to < 12 years (11 years, 364 days) at the time of consent
2. Confirmed clinical DSM-5 diagnosis of Autism Spectrum Disorder using the DSM-5 Checklist as informed by the Brief Observation of Symptoms of Autism (BOSA) and the Autism Diagnostic Interview-Revised (ADI-R)
3. Fragile X testing performed and negative; CMA and/or whole exome sequencing performed and results not linked to autism diagnosis
4. Stable on current psychiatric medication regimen (dose and dosing schedule) for at least 2 months prior to infusion of study product
5. Normal absolute lymphocyte count (≥1200/uL for African American participants and ≥1500/uL for all other participants)
6. GAI ≥ 65 via cognitive testing by study personnel
7. Participant and parent/guardian are English speaking
8. Able to travel to Duke University two times (baseline, six months), and parent/guardian is able to participate in interim surveys and interviews
9. Parental/guardian consent from at least one parent/guardian

Exclusion Criteria

1. General:

   1. Review of medical records and/or screening assessments indicates ASD diagnosis and/or GAI > 65 not confident
   2. Known diagnosis of any of the following coexisting psychiatric conditions: depression, bipolar disorder, schizophrenia, obsessive compulsive disorder associated with bipolar disorder, Tourette syndrome
   3. Screening data suggests that participant would not be able to comply with the requirements of the study procedures as assessed by the study team
   4. Family is unwilling or unable to commit to participation in all study-related assessments, including protocol follow up
   5. Sibling is enrolled in this (Duke IMPACT) study
2. Genetic:

   1. Records indicate that child has a known genetic syndrome such as (but not limited to) Fragile X syndrome, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cystic fibrosis, muscular dystrophy or a genetic defect definitively known to be associated with ASD
   2. Known pathogenic mutation or copy number variation (CNV) associated with ASD (e.g., 16p11.2, 15q13.2, 2q13.3)
3. Infectious:

   1. Known active CNS infection
   2. Evidence of uncontrolled infection based on records or clinical assessment
   3. Known HIV positivity
   4. Exposure to COVID-19 in the preceding 14 days or positive COVID-19 test in the previous 28 days. Subjects with a past history of infection with COVID-19 must be symptom-free for 14 days prior to the initial visit.
4. Medical:

   1. Known metabolic disorder
   2. Known mitochondrial dysfunction
   3. History of unstable epilepsy or uncontrolled seizure disorder, infantile spasms, Lennox Gastaut syndrome, Dravet syndrome, or other similar chronic seizure disorder
   4. Active malignancy or prior malignancy that was treated with chemotherapy
   5. History of a primary immunodeficiency disorder
   6. History of autoimmune cytopenias (i.e., ITP, AIHA)
   7. Coexisting medical condition that would place the child at increased risk for complications of study procedures
   8. Concurrent genetic or acquired disease or comorbidity(ies) that could require a future stem cell transplant
   9. Significant sensory (e.g., blindness, deafness, uncorrected hearing impairment) or motor (e.g., cerebral palsy) impairment
   10. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL or total bilirubin >1.3mg/dL, except in patients with known Gilbert's disease
   11. Significant hematologic abnormalities defined as: Hemoglobin <10.0 g/dL, Platelets <150 x 10e9/uL, WBC <3,000 cells/mL, ALC <1200/uL for African Americans or <1500/uL for all other participants.
   12. Evidence of clinically relevant physical dysmorphology indicative of a genetic syndrome as assessed by the PIs or other investigators, including a medical geneticist and psychiatrists trained in identifying dysmorphic features associated with neurodevelopmental conditions.
5. Current/Prior Therapy:

   a. Availability of a banked, qualified autologous cord blood unit or parents deferred use of qualified, autologous cord blood unit b. History of prior cell therapy c. Current or prior use of IVIG or other anti-inflammatory medications with the exception of NSAIDs d. Current or prior immunosuppressive therapy i. No systemic steroid therapy that has lasted >2 weeks, and no systemic steroids within 3 months prior to enrollment. Topical and inhaled steroids are permitted.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change on the Socialization and Communication Subscale Standard Scores on the Vineland Behavior Scales | Baseline, 6 months
  The primary outcome measure is the mean of the change on the Socialization and Communication Subscale Standard Scores on the Vineland Adaptive Behavior Scales (VABS-3). The primary endpoint is the change on this outcome measure from baseline to six months.

SECONDARY OUTCOMES:
Change in VABS-3 Socialization Standard Score | Baseline, 6 months
  Change in VABS-3 (Vineland Adaptive Behavior Scales) Socialization Standard Score
Change in VABS-3 Communication Standard Score | Baseline, 6 months
  Change in VABS-3 (Vineland Adaptive Behavior Scales) Communication Standard Score
Change in CGI-Severity score | Baseline, 6 months
  Clinical Global Impression- Severity Scale
CGI-Intervention score | Baseline, 6 months
  Clinical Global Impression- Impression
Change in the Pediatric Quality of Life Scale | Baseline, 6 months
  Pediatric Quality of Life Scale, raw scale range of 0-2300 with higher scores indicating a higher quality of life (better outcome)

OTHER OUTCOMES:
Incidence and severity of infusion reactions | Baseline, 6 months
  Assess for infusion reactions
Incidence and severity of product-related infections | Baseline, 6 months
  Assess for infections directly related to the study product infusions
Evidence of formation of anti-HLA antibodies | Baseline, 6 months, 12 months
  Assess for anti-HLA antibodies
Incidence and severity of graft versus host disease | 6 months, 12 months
  Assess for signs and symptoms of graft versus host disease
Incidence and severity of unexpected adverse events related to the study product | Baseline, 6 months, 12 months
  Assess for study related and unexpected adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Beth Shaz, MD, Principal Investigator — Duke University; Lauren Franz, MBChB, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No